CLINICAL TRIAL: NCT02442440
Title: Effectiveness of Anisodamine for the Treatment of Critically Ill Patients With Septic Shock: a Randomized Controlled Trial
Brief Title: Anisodamine Critically Ill SeptIc Shock
Acronym: ACIdoSIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, Zhongheng Zhang, Dr., Jinhua Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-013
Record Dates: First submitted 2015-04-30; First posted 2015-05-13 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock
Keywords: anisodamine; septic shock
MeSH Terms: conditions — Shock, Septic | interventions — anisodamine; 2-(phenylmethyl)-1-naphthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anisodamine group (Experimental): administration of the drug
  Interventions: Drug: anisodamine
- control group (No Intervention): these arm do not use anisodamine, other resuscitation protocol is as usual.

INTERVENTIONS:
Drug: anisodamine — Anisodamine will be given first as bolus of 10 mg, followed by 0.1-0.5mg/kg/hr. The adjustment of pump infusion rate is largely at the discretion of treating physician, with the aim of improving microcirculation and limit the side effect to a minimum. For example, if serum lactate continues to elevate, the infusion rate can be increased. Discontinuation on severe side effect or recovery of shock (normalized lactate, weaned from vasopressor) or death.
  Other Names: 654-2
  Arms: anisodamine group

SUMMARY:
Anisodamine has been widely used in China for its pharmacological effect on improving microcirculation during shock. It has been reported that anisodamine is effective in reducing mortality rate in children with meningitis. however, its effectiveness in patients with septic shock has not been systematically investigated. The aim of the study is to investigate the effectiveness of anisodamine in the treatment of patients with septic shock.

DETAILED DESCRIPTION:
Septic shock is an important contributor of mortality in the intensive care unit (ICU). The crude mortality is reported to be from 30% to 65% (1-5). Although there are significant advances in the management of septic shock in recent decades, the mortality rate was only marginally reduced. For example, the CUB-Réa Network study reported that the mortality rate of septic shock declined from 62.1% in 1993 to 55.9% in 2000 (6). The well-known Surviving Sepsis Campaign has also made every effort to reduce mortality rate of severe sepsis and septic shock. The organization recommended bundled strategies including early goal directed therapy (EGDT) for the management of septic shock (7,8). Although EGDT was once the mainstay therapy of septic shock, its efficacy has been questioned by recent several large randomized controlled trials (9,10). Therefore, the treatment of septic shock is still a global challenge and there is no well-established intervention that can reduce its mortality.

Anisodamine is an active agent isolated from a Chinese herb medicine. Both experimental and clinical studies have shown some potential beneficial effects of anisodamine in improving outcomes of shock (11-13). It was reported that anisodamine could reduce the mortality rate of fulminant epidemic meningitis from 66.9% to 12.4% (14). The efficacy of anisodamine might be mediated via the inhibition of thromboxane synthesis, granulocyte and platelet aggregation (15). Although anisodamine has been widely used in the treatment of septic shock in mainland China, there is no solid evidence from well designed clinical trials to support its efficacy. The aim of the study is to investigate the effectiveness of anisodamine in the treatment of critically ill patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* patients with septic shock

Inclusion criteria included patients with sepsis plus use of vasopressors. Systemic inflammatory response syndrome (SIRS) is defined as meeting at least one of the following 3 criteria for a systemic inflammatory response. One of the SIRS criteria must be either the WBC criteria (a) or the body temperature criteria (b):

1. White blood cell count >12,000 or <4,000 or >10% band forms
2. Body temperature >38oC (any route) or <36oC (accepting core temperatures only; indwelling catheter, esophageal, rectal)
3. Heart rate (> 90 beats/min) or receiving medications that slow heart rate or paced rhythm.

Suspected or documented infection included the following sites: thorax, urinary tract, abdomen, skin, sinuses, central venous catheters, and bacterial meningitis.

Septic shock was defined as sustained arterial hypotension with systolic blood pressure (SBP) < 90 mm Hg, mean arterial pressure (MAP) < 70 mm Hg, or an SBP decrease > 40 mm Hg, despite adequate fluid resuscitation. To ease clinical screening process, we defined septic shock as the requirement of vasopressors despite adequate fluid resuscitation. Vasopressors include norepinephrine, epinephrine, phenylephrine and dopamine>5mcg/kg/min.

Patients with following conditions will be excluded:

1. Age<15 years old
2. Moribund (expected to die within 24 hours)
3. Stay in ICU for more than 24 hours
4. Contraindications to anisodamine: elevated intracranial pressure, acute phase of intracranial hemorrhage, glaucoma, untreated bowel obstruction (surgically treated obstruction is not contraindicated), enlargement of prostate without urinary catheterization.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2015-04; Primary Completion 2020-10 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
hospital mortality | from ICU admission to hospital discharge (participants will be followed for the duration of hospital stay, an expected average of 28 days)
  the outcome will be assessed by using proportion of patients died, and relative risk will be reported.

SECONDARY OUTCOMES:
lactate levels | from ICU admission to hospital discharge (participants will be followed for the duration of hospital stay, an expected average of 28 days)
  the value was measured in mmol/l, and they will be compared between both arms.

CONTACTS AND LOCATIONS:
Overall Officials: kun chen, MSc, Study Director — Jinhua Municipal Central Hospital
Locations (14):
- China (14):
  - Huizhou first hospital, Huizhou, Guangdong
  - Union Hospital, Tongji medical collegue, Huazhong university of Science and Technology, Wuhan, Hubei
  - the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - affiliated hospital, Jiangsu University, Zhenjiang, Jiangsu
  - Binzhou People's hospital of Shandong province, Binzhou, Shandong
  - department of critical care medicine, Ren Ji Hospital, School of medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Peace hospital of Changzhi medical college, Changzhi, Shanxi
  - The first People's hospital of Yongkang, Guli, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw hospital, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Department of critical care medicine, The central hospital of Lishui City, Lishui, Zhejiang
  - Beilun People's hospital; The first affiliated hospital of Zhejiang university (Beilun Branch), Ningbo, Zhejiang
  - Taizhou hospital of Zhejiang province, Taizhou, Zhejiang

REFERENCES:
- [Derived] Yu Y, Zhu C, Hong Y, Chen L, Huang Z, Zhou J, Tian X, Liu D, Ren B, Zhang C, Hu C, Wang X, Yin R, Gao Y, Zhang Z. Effectiveness of anisodamine for the treatment of critically ill patients with septic shock: a multicentre randomized controlled trial. Crit Care. 2021 Sep 27;25(1):349. doi: 10.1186/s13054-021-03774-4. PMID 34579741
- [Derived] Zheng Y, Li Y, Liu X, Zhang R, Wang Z, Sun H, Liu S. A phase III, multicenter randomized controlled trial of neo-adjuvant chemotherapy paclitaxel plus cisplatin versus surgery alone for stage IIA-IIIB esophageal squamous cell carcinoma. J Thorac Dis. 2017 Jan;9(1):200-204. doi: 10.21037/jtd.2017.01.44. PMID 28203424
- [Derived] Zhang Z, Zhou J, Shang Y, Wang X, Yin R, Zhu Z, Chen W, Tian X, Yu Y, Zuo X, Chen K, Ji X, Ni H; Anisodamine Critically Ill SeptIc Shock (ACIdoSIS) study group. Effectiveness of anisodamine for the treatment of critically ill patients with septic shock (ACIdoSIS study): study protocol for randomized controlled trial. Ann Transl Med. 2015 Oct;3(17):246. doi: 10.3978/j.issn.2305-5839.2015.10.03. PMID 26605292